CLINICAL TRIAL: NCT04329416
Title: Efficacy of Height-Based Formula to Predict Insertion Depth of Left-Sided Double Lumen Tube. A Prospective Observational Study
Brief Title: Insertion Depth of Left-sided Double-lumen Tube: a New Predictive Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: King Saud University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E-18-3064
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Thoracic Surgery; One Lung Ventilation; Left-sided Double Lumen Tube

STUDY DESIGN:
Intervention Model Description: A prospective observational single-center open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Predicted depth of insertion (Other): The predicted insertion depth of the DLT was calculated using the formula [0.249 x (BH) 0.916] before induction of anesthesia using an application on the smartphone
  Interventions: Other: Predicted depth of insertion; Other: Optimized depth of insertion; Other: Adjustment of depth of insertion

INTERVENTIONS:
Other: Predicted depth of insertion — A left-sided double-lumen tube was introduced beyond the vocal cords when the train-of-four stimulation of the ulnar nerve revealed 1 or 2 twitches, the stylet was removed, the double-lumen tube was rotated 90° counterclockwise and then advanced blindly to the predicted depth of insertion.
Other: Optimized depth of insertion — The optimal position of the double-lumen tube, defined as the inflated endobronchial cuff is placed in the left main bronchus just below the carina without herniation, which was confirmed using a flexible bronchoscope in both supine and lateral decubitus positions.
Other: Adjustment of depth of insertion — If the endobronchial cuff was placed too deeply or too proximal, subsequently, the double-lumen tube was withdrawn or advanced, respectively, using the flexible bronchoscope until the optimum position of the double-lumen tube was achieved.

SUMMARY:
The authors developed a formula for predicting the accurate depth of DLT insertion into the appropriate bronchus based on height as follows [The predicted insertion depth of left DLT (cm) equals 0.249 × (BH)0.916] [R]. That pilot study showed comparable correlations between five formulae [Brodsky et al, Bahk and Oh R, Takita et al, Chow et al, Lin]. However, that formula developed has not been validated yet.

We hypothesized that previously published formula would predict the accurate depth of left-sided DLT insertion. We aimed to investigate the efficacy of this formula to estimate the optimum insertion depth of the DLT using a flexible bronchoscope and decrease the incidence of DLT displacement into the appropriate bronchus, the need for bronchoscopic adjustment, and complications including soreness of throat and mucosal injury.

DETAILED DESCRIPTION:
Accurate placement of the double-lumen tube [DLT], the commonly used tool to provide one-lung ventilation during thoracic surgery, is a real challenge for the thoracic anesthesiologists. Optimal DLT depth, defined as the blue endobronchial cuff below the carina, would decrease the incidence of obstructing the trachea and the contralateral bronchus (Brodsky). Additionally, deep insertion of the bronchial cuff of the DLT would obstruct the upper lobe bronchus (Brodsky). The careful adjustment of the depth and optimal positioning of the DLT using a flexible fiberoptic bronchoscope need a skilled anesthesiologist to reduce the time to DLT intubation. (Charles D. Boucek et al)

There are several methods have been described to predict the proper depth of DLT insertion. Chow et al. documented the validity of the developed formula based on the clavicular-to-carinal distance of trachea and height in 78% of patients studied. Brodsky et al. demonstrated that a height-and-gender-based formula could predict the depth of DLT insertion. Liu et al. reported an accurate depth of DLT insertion in 90% of patients studied measuring the distance between the vocal cord and carina according to the chest CT.

ELIGIBILITY:
Inclusion Criteria:

* Underwent thoracic surgery
* Using a left-sided double-lumen tube for one-lung ventilation

Exclusion Criteria:

* Anticipated or known difficult airway
* Refuse to sign the consent
* Withdraw the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
The rate of optimum position of the double-lumen tube | for 15 minutes after double-lumen tube insertion
  The rate of optimum position of a left-sided DLT without further adjustments, defined as the inflated endobronchial cuff is placed in the left main bronchus just below the carina without herniation

SECONDARY OUTCOMES:
The calculated predicted depth of insertion | immediately before induction of general anesthesia
  The predicted insertion depth of the DLT was calculated using the formula [0.249 x (BH) 0.916] using an application an application on the smart phone
The initial depth of insertion | for 15 minutes after double-lumen tube insertion
  The "initial depth of insertion," was measured using the external centimeter markings on the DLT's lumen at the level of incisors
Position of the double-lumen tube with the flexible bronchoscope | for 15 minutes after double-lumen tube insertion
  The position of the DLT with the flexible bronchoscope would be rated either (1) optimally placed, (2) too far out, or (3) too far in
The need for bronchoscopic adjustments | for 15 minutes after double-lumen tube insertion
  If the endobronchial cuff was placed too deeply or too proximal, subsequently, the DLT was withdrawn or advanced, respectively, using the flexible bronchoscope until the optimum position of the DLT was achieved. The optimizing maneuvers were recorded
The final correct depth of insertion | for 15 minutes after double-lumen tube insertion
  the "final correct depth of insertion", defined as the distance from the distal opening of the bronchial lumen to the corner of the mouth, was measured with a flexible bronchoscope passing through the bronchial lume
Time to final correct double-lumen tube positioning | for 25 minutes after double-lumen tube insertion
  Time to final correct DLT positioning from time of laryngoscopy was recorded
Changes in heart rate | for 25 minutes after double-lumen tube insertion
  Postintubation changes in heart rate was recorded
Changes in mean arterial blood pressure | for 25 minutes after double-lumen tube insertion
  Postintubation changes in mean arterial blood pressure was recorded
Changes in peripheral oxygen saturation | for 25 minutes after double-lumen tube insertion
  Postintubation changes in peripheral oxygen saturation was recorded
Degree of lung collapse | for 30 minutes after start of surgery
  degree of lung collapse was rated as excellent, good, poor, or very poor
The incidence of soreness of throat | for 24 hours after start of surgery
  Patients were asked about the occurrence and severity of postoperative sore throat
The incidence of mucosal injury | for 40 minutes after double-lumen tube insertion
  The incidence of mucosal injury using the flexible bronchoscope was reported after intubation using the double-lumen tube

CONTACTS AND LOCATIONS:
Overall Officials: Abdelazeem A Eldawlatly, MD, Study Chair — Professor of Anesthesia, College of Medicine, King Saud University; Mohamed R El Tahan, MD, Study Director — Associate Professor of Cardiothoracic Anaesthesia & Surgical Intensive Care, Imam Abdulrahman Bin Faisal University (formerly, University of Dammam), Dammam, Saudi Arabia,
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, the anonymized database would be shared after publishing the paper
Supporting Information: Study Protocol, SAP
Time Frame: Unlimited time starting after publishing the paper